CLINICAL TRIAL: NCT00639379
Title: A Multi-Center, Subject Masked, Randomized, Two Week Crossover Design, Investigation of the Acuvue Cypress Toric Silicone Hydrogel Lens Compared to the Bausch & Lomb SofLens66® Toric Hydrophilic Lens
Brief Title: Comparison of Two Toric Contact Lenses on Current Toric Wearers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CR-0802
Record Dates: First submitted 2008-03-13; First posted 2008-03-20 (Estimated); Results first posted 2010-07-19 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Ametropia
Keywords: toric contact lenses; vision; comfort; toric fit characteristics; slit lamp findings
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- senofilcon A (Experimental): senofilcon A toric daily wear contact lenses
  Interventions: Device: senofilcon A toric
- alphafilcon A (Active Comparator): alphafilcon A toric daily wear contact lenses
  Interventions: Device: alphafilcon A toric

INTERVENTIONS:
Device: senofilcon A toric — silicone hydrogel toric lens, 2 wk replacement, daily wear
  Other Names: ACUVUE OASYS
  Arms: senofilcon A
Device: alphafilcon A toric — hydrogel toric lens, 2 wk replacement, daily wear
  Other Names: SofLens Toric
  Arms: alphafilcon A

SUMMARY:
The purpose of this study is to evaluate and compare the clinical performance of two toric contact lenses amongst 110 subjects, 2-week, single masked (subject), daily wear, randomized, bilateral, crossover study; 4 weeks duration. Hypotheses include equal or better performance of the test lens over the control lenses for comfort, vision, and toric fit characteristics as well as corneal integrity

DETAILED DESCRIPTION:
Up to 7 sites in the US will participate. Each investigator will have both test and control lens types. There will be a maximum of 6 scheduled visits:

Visit 1: Habitual lens evaluation / Baseline / Trial fitting Visit 2: Dispensing (to be combined with Visit 1 where possible), Visit 3: Questionnaire only (no exam) 7 days (±2) after dispensing, Visit 4: 2 week follow-up 14 days (±3) after dispensing, and dispense second lens type, Visit 5: Questionnaire only (no exam) 7 days (±2) after 2nd lens dispense, Visit 6: 2 week follow-up 14 days (±3) after 2nd lens dispense

ELIGIBILITY:
Inclusion Criteria:

1. Be at least 18 and less than or equal to 45 years of age, have a need for vision correction and wear contact lenses in BOTH eyes (monovision or uni-ocular fitting is NOT allowed).
2. Be able to read J1 at near WITHOUT the aid of a near addition over the distance prescription.
3. Be a currently successful wearer for at least 3 months of B&L SofLens 66 Toric hydrogel lenses.
4. Be able and willing to adhere to the instructions set forth in the protocol.
5. Agree to wear their contact lenses in both eyes on a daily wear schedule for at least 8 hours per day every day during the study.
6. Have a distance spectacle spherical component between -1.00 D and -5.25 D with cylinder in the range of 0.75 D to 2.25 D and cylinder axis within 10 ° of the vertical and within 30° of the horizontal in both eyes (when the subject's prescription is presented in minus cylinder form).
7. Have a best corrected manifest refraction visual acuity of at least 20/25 or better in each eye.
8. Be in good general health, based on his/her knowledge.
9. Must be given an explanation of the study objectives, lens and solutions usage requirements and visit schedule. The subject must read, indicate understanding of and agree to begin participation in the clinical study. The subject must then sign the Informed Consent Form in the presence of the Investigator or their designee.

Exclusion Criteria:

1. Presbyopic or has the need for a near add for reading.
2. Previous refractive surgery; current or previous orthokeratology treatment.
3. Aphakia, keratoconus or a highly irregular cornea.
4. The presence of ocular or systemic disease or has the need for medication (ocular or systemic) which might interfere with contact lens wear or which would cause the lenses to be removed more than twice a day. (e.g., Sjögren's syndrome, type II diabetes, allergies).
5. A known history of corneal hypoesthesia (reduced corneal sensitivity.)
6. Anterior uveitis or iritis (past or present).
7. A history of recurrent erosions, corneal infiltrates corneal ulcer or fungal infections.
8. Clinically significant (grade 3 or 4) anterior segment abnormalities; inflammations or infections of the eye, eyelids, or associated structures.
9. Slit lamp findings that would contraindicate contact lens wear such as:

   * Pathological dry eye or associated findings
   * Pterygium or corneal scars within the visual axis
   * Neovascularization >1mm in from the limbus
   * History of giant papillary conjunctivitis (GPC) worse than Grade 2
   * Meibomian gland dysfunction, blepharitis, or seborrhoeic dermatitis
10. Current pregnancy or lactation (to the best of the subject's knowledge).
11. Actively participating in another clinical study at any time during this study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 89 (Actual)
Dates: Start 2008-02; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Ted Brink and Associates, Jacksonville, Florida
  - Eola Eyes, Orlando, Florida
  - Clayton Eye Center, Morrow, Georgia
  - The Koetting Associates Inc., St Louis, Missouri
  - Southern Eyes, Concord, North Carolina
  - Western Reserve Vision Care, Beachwood, Ohio
  - Primary Eyecare Group, P.C., Brentwood, Tennessee

RESULTS

PARTICIPANT FLOW:
Groups:
- Senofilcon A Toric / Alphafilcon A Toric: senofilcon A toric work bilaterally during first 2-week period, alphafilcon A toric work bilaterally during second 2-week period.
- Alphafilcon A Toric / Senofilcon A Toric: alphafilcon A toric work bilaterally during first 2-week period, senofilcon A toric work bilaterally during second 2-week period.
Period: Period 1 - 2 Weeks
Arm/Group | Senofilcon A Toric / Alphafilcon A Toric | Alphafilcon A Toric / Senofilcon A Toric
Started | 44 | 45
Completed | 39 | 45
Not Completed | 5 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — lens issue | 3 | 0
Period: Period 2 - 2 Weeks
Arm/Group | Senofilcon A Toric / Alphafilcon A Toric | Alphafilcon A Toric / Senofilcon A Toric
Started | 39 | 45
Completed | 39 | 45
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Total Completed Participants
Number analyzed (Participants) | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.6 (8.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53
  Male | 31

OUTCOME MEASURES:

1. Primary Outcome: Lens Orientation Within 5 Degrees
Description: Number of eyes with lens orientation within 5 degrees of optimal orientation within 1 minute of contact lens insertion.
Time Frame: 1 minute after insertion
Population: Subjects/eyes that completed the study were analyzed. A total of 168 eyes/84 subjects were analyzed.
Measure: Number; unit: Eyes
Arm/Group | Senofilcon A Toric | Alphafilcon A Toric
Number analyzed (Participants) | 84 | 84
Eyes | 128 | 128
Statistical Analysis 1: Comparison: Senofilcon A Toric vs Alphafilcon A Toric; Alternative hypothesis is that senofilcon A toric is non-inferior to alphafilcon A toric for proportion of eyes with lens orientation within 5 degrees; Test type: Non-Inferiority or Equivalence — Non-inferiority margin is 0.65; Regression, Logistic; Odds Ratio (OR) = 0.967, 98.98% CI 2-sided [0.436 to 0.967] — Odds ratio is senofilcon A toric / alphafilcon A toric

2. Primary Outcome: Lens Stability
Description: Number of eyes with the amount of rotation induced from a blink within 5 degrees of settled orientation.
Time Frame: 10-15 minutes after insertion
Population: Subjects/eyes that completed the study were analyzed. A total of 168 eyes/84 subjects were analyzed.
Measure: Number; unit: Eyes
Arm/Group | Senofilcon A Toric | Alphafilcon A Toric
Number analyzed (Participants) | 84 | 84
Eyes | 144 | 138
Statistical Analysis 1: Comparison: Senofilcon A Toric vs Alphafilcon A Toric; Alternative hypothesis is that senofilcon A toric is non-inferior to alphafilcon A toric for proportion of eyes with lens stability within 5 degrees; Test type: Non-Inferiority or Equivalence — Non-inferiority margin = 0.65; Regression, Logistic; Odds Ratio (OR) = 1.416, 98.98% CI 2-sided [0.680 to 1.416] — Odds ratio is senofilcon A toric / alphafilcon A toric

3. Primary Outcome: Subjective Lens Comfort
Description: A weighted combined score calculated from individual comfort-related questions asked on a 1-5 scale: 1=most negative response to 5=most positive response, was used to derive comfort outcomes. The analysis shows the difference in outcome between the test and control. >0=comfortable, <0=uncomfortable.
Time Frame: 1 and 2 weeks
Population: Subjects that completed the study were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Senofilcon A Toric | Alphafilcon A Toric
Number analyzed (Participants) | 84 | 84
Units on a scale | 0.08125 (0.08771) | -0.1055 (0.08771)
Statistical Analysis 1: Comparison: Senofilcon A Toric vs Alphafilcon A Toric; Alternative hypothesis is that senofilcon A toric is non-inferior to alphafilcon A toric for lens comfort; Test type: Non-Inferiority or Equivalence — Non-inferiority margin = -0.4; Mixed Models Analysis; Mean Difference (Final Values) = 0.1868, 98.98% CI 2-sided [-0.0517 to 0.1868], Standard Error of Mean 0.0921 — The mean difference is calculated as senofilcon A toric minus alphafilcon A toric

4. Primary Outcome: Subjective Vision
Description: A weighted combined score calculated from individual vision-related questions asked on a 1-5 scale: 1=most negative response to 5=most positive response, was used to derive vision outcomes. The analysis shows the difference in outcome between the test and control. >0=satisfactory vision, <0=unsatisfactory vision.
Time Frame: 1 and 2 weeks
Population: Subjects that completed the study were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Senofilcon A Toric | Alphafilcon A Toric
Number analyzed (Participants) | 84 | 84
Units on a scale | -0.0420 (0.08885) | -0.0302 (0.08885)
Statistical Analysis 1: Comparison: Senofilcon A Toric vs Alphafilcon A Toric; Alternative hypothesis is that senofilcon A toric is non-inferior to alphafilcon A toric for subjective vision; Test type: Non-Inferiority or Equivalence — Non-inferiority margin = -0.4; Mixed Models Analysis; Mean Difference (Final Values) = -0.01185, 98.98% CI 2-sided [-0.2337 to -0.01185], Standard Error of Mean 0.08566 — The mean difference is calculated as senofilcon A toric minus alphafilcon A toric

5. Primary Outcome: Overall Corneal Staining
Description: Corneal staining measured using the National Eye Institute grading scale of grade 0 = normal, grade 1 = mild, grade 2 = moderate, grade 3 = severe.
Time Frame: after 2 weeks use
Population: Subjects that completed the study were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Senofilcon A Toric | Alphafilcon A Toric
Number analyzed (Participants) | 84 | 84
Units on a scale | 0.04921 (0.01174) | 0.06188 (0.01176)
Statistical Analysis 1: Comparison: Senofilcon A Toric vs Alphafilcon A Toric; Alternative hypothesis is senofilcon A toric is non-inferior to alphafilcon A toric by having a lower level of corneal staining; Test type: Non-Inferiority or Equivalence — Non-inferiority margin = 0.5; Mean Difference (Final Values) = -0.01267, 98.98% CI 2-sided [-0.01267 to 0.01986], Standard Error of Mean 0.01265 — The mean difference was calculated as senofilcon A toric minus alphafilcon A toric

ADVERSE EVENTS:
Arm/Group | Senofilcon A Toric / Alphafilcon A Toric | Alphafilcon A Toric / Senofilcon A Toric
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/45
Other Adverse Events (participants affected / at risk) | 0/44 | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI may not publish, divulge, reveal, disclose, or use the data and or results of the study without prior written consent of Vistakon.